CLINICAL TRIAL: NCT01557153
Title: Vascular Augmentation of Late-life Unremitted Depression (VALUeD)
Acronym: VALUeD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gateshead Health NHS Foundation Trust (Other)
Collaborators: Newcastle-upon-Tyne Hospitals NHS Trust (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 724; RfPB PB-PG-0609-19028 (Other Grant/Funding Number: NIHR RfPB); 2010-023969-21 (EudraCT Number)
Record Dates: First submitted 2012-03-13; First posted 2012-03-19 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Depression
Keywords: Late-life Unremitted Depression
MeSH Terms: conditions — Depression | interventions — Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amlodipine (Experimental)
  Interventions: Drug: Amlodipine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amlodipine — Starting dose will be 5mg/day for four weeks. All participants will be titrated up to the maximum of 10mg/day after 4 weeks. If they do not tolerate this dose, it will be reduced again to 5mg/day and they will continue on their maximum tolerated dose for 12 weeks (for a total of 16 weeks of medication or placebo)
  Arms: Amlodipine
Drug: Placebo — Starting dose will be 5mg/day for four weeks. All participants will be titrated up to the maximum of 10mg/day after 4 weeks. If they do not tolerate this dose, it will be reduced again to 5mg/day and they will continue on their maximum tolerated dose for 12 weeks (for a total of 16 weeks of medication or placebo)
  Arms: Placebo

SUMMARY:
Depression has a high occurrence and causes other problems in older people, two thirds of these patients will not have a lessening in their condition from routine treatment medication. About half have a form of depression known as 'vascular depression'. Augmentation, the addition to, antidepressant treatment with a vascular type of treatment (such as a group of medications called Calcium Channel Blocker including the medication called amlodipine) may be effective in this group of patients but previously published studies have been from highly selected specific patient groups. The investigators would like to find out if giving amlodipine medication to people with late life non-responding vascular depression would be acceptable to this patient group. The investigators would also like to know how they feel while having the treatment and whether this provides a measurable benefit for those patients and whether those benefits are relevant to the patients. The investigators would also like to find out the information the investigators need to plan and prepare for a larger version of this study.

DETAILED DESCRIPTION:
Depression has a high prevalence and causes other problems in older people. Two-thirds of these patients will not have an improvement in their condition from routine treatment. About hald have a form of depression known as 'Vascular Depression'. Augmentation, in this case the addition to antidepressant treatment of a vascular type of treatment (such as a group of medications called Calcium Channel Blockers including the medication called amlodipine) may be effective in this group of patients but previously published studies have been from highly selected specific patient groups. We would like to find out if giving amlodipine medication to people with late life non-responding vascular depression would be acceptable to this patient group. We would also like to know how they feel while having the treatment and whether this provides a measureable benefit for those patients and whether those benefits are relevant to the patients. We would also like to find out the information we need to plan and prepare for a larger version of this study.

Participants may be eligible for the study if they are 50 years old or over, and have been diagnosed with depression which has not gotten better with other drugs, we call this type of depression 'Vascular Depression'.

If a participant would like to be involved in this study, they would be required to attend the Clinical Ageing Research Unit (CARU) at the former Newcastle General Hospital site in Newcastle upon Tyne for up to seven visits as part of this clinical trial, and would be required to take the study medication prescribed to them. The study medication may be either amlodipine or placebo, however neither the participant nor the doctor or nurses involved in the study will be aware of which medication has been given. This is called a double blind study, and is done to ensure that there is no other influence on the results apart from the effects of the drug itself. Each participant will be randomly assigned to receiving either amlodipine or placebo in a process called randomisation.

As part of this study, participants will be invited to attend the unit mentioned above for their study visit, the first of which will be to discuss this study in further detail and allowing the participant time to ask any questions and to consider their participation in the study. If they would like to be involved, they will be invited to return for a second visit at which time they will be asked to give their consent to be involved in the study. They will then need to have their blood pressure taken, have an ECG (electrocardiograph) to establish how well their heart is working, have a small blood sample taken and complete four short questionnaires.

Following on from this, the participant will be invited back for another visit, which will also be used to confirm the participants eligibility. At this visit the participant will be required to have a physical examination from the study doctor, have their blood pressure checked and complete the nine short questionnaires. Once a participant has been confirmed as eligible for the study, they will be entered into the study and randomised to receive either amlodipine or placebo. The participant will then receive four weeks supply of the study medication.

Two weeks after this visit, and again at 6 weeks and 12 weeks into the study, each participant will be contacted by the research study nurses in order to review how the participant has been since their last visit.

At weeks 4 and 8 of the study, participants will be required to attend the research centre for another visit at which point they will be asked to complete two short questionnaires, have their blood pressure taken and current medication reviewed, and will receive their next supply of study medication.

At 16 weeks after starting the study, study medication will be stopped and participants will be asked to attend another visit at which time current medication will be reviewed, blood pressure will be assessed, as well as a blood sample will be taken. Participants will also be asked to complete eight short questionnaires. Depending on the results of these questionnaires, participants may be asked to attend for another visit a week later at which point their blood pressure will be taken again, and they will be asked to complete six short questionnaires.

At 20 weeks after the start of the study, patients will be asked to return for a final visit at which point they will be asked to complete two short questionnaires and have their blood pressure taken once more.

Following on from this study, participants will be returned to the care of their GP.

As part of this study, participants will also be invited to take part in an interview, which will involve the discussion of the various questionnaires undertaken in the study and any other concerns the participant may have had during the course of the study. These interviews will be optional and not be a required part of the study, should the participant decline to take part in the interviews they will still be able to remain in the main part of the study.

There is no guarantee that taking part in this study may benefit the participant, however it is anticipated that the active medication could reduce the symptoms of their depression. The risk involved in participating in this study is very small, and may include the small risk of bruising or infection at the site where the blood sample was taken. Other risks include the possible side effects of the study drug (amlodipine) which may include swelling of the ankles, dizziness, fatigue, nausea, indigestion, palpitations or headaches. These, and other side effects, are listed in the Patient Information sheet which will be given to each potential participant for further information.

Potential participants will be identified at their GP practices which will be involved in the study as Participant Identification Centres (PICs).

The study is being sponsored by Gateshead Health NHS Foundation Trust, and is funded by the National Institute for Health Research - Research for Patient Benefit. The study will start around the 1st April 2012 and will run for approximately 24 months.

The main contact for any potential participant for this study will be Julie Henry (Research Nurse) based at the Clinical Ageing Research Unit, Campus for Ageing and Vitality, Newcastle upon Tyne, NE4 5PL, Telephone: 0191 248 1280 (reception)

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years or more
* Clinically significant (unremitted) vascular depression, as defined above.
* MMSE > 23
* BP < 150/90 (QoF Audit standard)
* Patient has provided written informed consent for participation in the study prior to any study specific procedures

Exclusion Criteria:

* Taking a calcium channel blocker
* Clinical evidence of dementia
* History or clinical evidence of stroke
* History of bipolar or psychotic disorder
* Significant suicide risk
* Known hypersensitivity to amlodipine or any other calcium channel blocker
* Severe renal or hepatic impairment
* Pregnancy, or women planning to become pregnant within next 12 months, or women who are breast feeding
* Use of other investigational study drugs within 30 days prior to study entry (defined as date of randomisation into study)
* Presence of cardiac pace-maker or other contraindications to (only applied to those consenting MRI sub-study)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-04; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Response rates to study invitation to GP practices and patients | 24 months
  To determine the response rates to study invitiation by GP practices (for involvement as a PIC) and patients (for study participation)

SECONDARY OUTCOMES:
HAM-D score of less than 10 for 2 consecutive assessments | 16 weeks
  To measure remission (HAM-D < 10 for 2 consecutive assessments) by 16 weeks of augmentation
Ham-D reduction in symptoms | 16 weeks
  To review any reduction in symptoms over the 16 weeks treatment period as shown by the HAM-D questionnaire
Geriatric Depression Scale questionnaire | 16 weeks
  to measure and record responses and changes reported on the GDS questionnaire over the course of treatment
EQ-5D questionnaire | 16 weeks
  To review reponses and changes in responses to the EQ-5D over the course of 16 weeks of treatment
Clinical Global Impression severity and improvement | 16 weeks
  The CGI questionnaires will be reviewed for severity and any improvement over the course of the 16 week treatment
Instrumental Activities of Daily Living questionnaire | 16 weeks
  to review reponses and changes reported in the IADL questionnaire over the course of 16 weeks of treatment
reduction in symptoms (HAM-D) in those with significant baseline white matter hyperintensities | 16 weeks
  To review any reduction in symptoms on the HAM-D questionnaire over the course of 16 weeks in participants with significant WMH as shown on MRI scan
Blood pressure | 16 weeks
  To review blood presure in participants over the course of 16 weeks of treatment
Effect of treatment on perfusion | 16 weeks
  to evaluate the effect of treatment on perfusion as determine by second MRI scan

CONTACTS AND LOCATIONS:
Overall Officials: Alan Thomas, Dr, Principal Investigator — Gateshead Health NHS Foundation Trust
Locations (1):
- Clinical Ageing Research Unit, Newcastle upon Tyne, United Kingdom